CLINICAL TRIAL: NCT06413732
Title: The Effect of Dual Task Training on Gait, Balance, and Quality of Life in Patients With Stroke
Brief Title: The Effect of Dual Task Training in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Tarik Ozmen, Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Karabuk Physiotherapy
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): The dual-task training program combined with conventional physiotherapy was applied to both groups for approximately 1 hour, 5 days a week.
  Interventions: Other: Conventional physiotherapy
- Group II (Other): Only conventional physiotherapy was applied to both groups for approximately 1 hour, 5 days a week.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Conventional physiotherapy — Conventional physiotherapy was applied for approximately 1 hour, 5 days a week.

SUMMARY:
The aim of this study was to investigate the effect of dual-task training on gait, balance, and quality of life in individuals with stroke. The study included 30 individuals aged 30-80 years with stroke. All participants were assessed using the 10-meter walk test (10MWT), 10MWT under dual-task interaction (DTI), timed up and go (TUG), 30-Second Chair-Stand Test (30s-CST), Berg Balance Scale (BBS), Short Form 36 (SF-36). Participants were randomized into two groups. Both groups received conventional physiotherapy for approximately 1 hour, five days a week. Group I also received dual-task training.

ELIGIBILITY:
Inclusion Criteria:

* Having a score of 24 or above on the Mini-Mental State Test,
* Being able to walk at least 10 meters without using a walking aid
* Having a total score of 5 on the motor and cognitive sections of the Functional Independence Scale.

Exclusion Criteria:

* Neurological and orthopedic problems that could affect motor performance and balance
* Communication problems
* Patients who had received Botulinum Toxin injection treatment in the last six months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Six weeks
  It is a scale designed to evaluate balance and determine the risk of falling. It consists of 14 items based on performance of sitting, standing, and posture change. Scores can range from 0 to 56. The higher the score, the better the postural control.
Timed Up and Go Test | Six weeks
  The participant was asked to get up from the chair he was sitting on, walk 3 meters at a safe and normal speed, and then turn back and sit on the chair again. The time was recorded by a stopwatch.
10-meter walk test | Six weeks
  The 10-meter walk test (10MWT) is suggested for assessing gait in post-stroke rehabilitation. The participant was instructed to walk at comfortable walking speed a distance of 10 meters. The time was recorded in seconds with a stopwatch.
30-Second Chair-Stand Test | Six weeks
  For this test, the participant was seated on a chair with a sitting height of 45-47 cm, with his arms on his chest, and was asked to stand up and sit down as many times as possible within 30 seconds. The score was recorded as zero if the participant could not get up from the chair without using their arms
Short Form 36 | Six weeks
  The scale consists of 36 items in the following categories: physical function, social function, physical role, emotional role, mental health, vitality, bodily pain, and general health. Subscales evaluate health between 0 and 100, with 0 indicating poor health and 100 indicating good health.
  The scale consists of 36 items in the following categories: physical function, social function, physical role, emotional role, mental health, vitality, bodily pain, and general health. Subscales evaluate health between 0 and 100, with 0 indicating poor health and 100 indicating good health.
  The scale consists of 36 items in the following categories: physical function, social function, physical role, emotional role, mental health, vitality, bodily pain, and general health. Subscales evaluate health between 0 and 100, with 0 indicating poor health and 100 indicating good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarik Ozmen, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No